CLINICAL TRIAL: NCT01322620
Title: Haemophilia, Experiences, Results and Opportunities (HERO): A Community-based Evaluation of the Psychosocial Effects of Haemophilia on Patients and Their Carers
Brief Title: Survey Evaluating the Psychosocial Effects of Living With Haemophilia
Acronym: HERO
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-3911; U1111-1119-7128 (Other: WHO)
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors; Relatives to/Carers of Patients
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given. Participants are to complete a questionnarie in the study.

SUMMARY:
This study is conducted in Africa, Asia, Europe, North America and South America.

The purpose of the survey is to identify the key psychosocial issues affecting patients with haemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Males with haemophilia A or B (with or without inhibitors)
* Parents/carers of children aged below 18 years with haemophilia A or B (with or without inhibitors)
* Patients currently receiving treatment for haemophilia with one of the following: replacement factor VIII or replacement factor IX or a bypassing agent (recombinant factor VIIa or aPCC (Activated prothrombin complex concentrate))
* Patients with haemophilia, not currently receiving treatment with replacement factor VIII or IX or a bypassing agent (as appropriate), but who have had at least one spontaneous bleed into one or more joints within the last 12 months
* Subjects must have access to the internet, either at home or at a location convenient to them, be able to complete a paper questionnaire, or be available to attend a face-to-face interview (Algerian subjects only), to participate in the survey

Exclusion Criteria:

* Inability to understand and comply with written and verbal instructions unless assisted at the haemophilia treatment centre (HTC) or by a relative

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males with haemophilia and parents/carers of children with haemophilia.
Sampling Method: Non-Probability Sample
Enrollment: 1236 (Actual)
Dates: Start 2011-06-03 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2012-02-29 (Actual)

PRIMARY OUTCOMES:
To quantify the extent of key psychosocial factors affecting patients with haemophilia in their daily lives | After 6 weeks (recruitment and data collection)

SECONDARY OUTCOMES:
To quantify how psychosocial factors are associated with treatment outcomes, compliance, health and general well-being | After 6 weeks (recruitment and data collection)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Novo Nordisk Investigational Site, Mississauga, Canada
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Crawley, United Kingdom

REFERENCES:
- [Result] Forsyth AL, Gregory M, Nugent D, Garrido C, Pilgaard T, Cooper DL, Iorio A. Haemophilia Experiences, Results and Opportunities (HERO) Study: survey methodology and population demographics. Haemophilia. 2014 Jan;20(1):44-51. doi: 10.1111/hae.12239. Epub 2013 Aug 1. PMID 23902228
- [Result] Witkop M, Guelcher C, Forsyth A, Hawk S, Curtis R, Kelley L, Frick N, Rice M, Rosu G, Cooper DL. Treatment outcomes, quality of life, and impact of hemophilia on young adults (aged 18-30 years) with hemophilia. Am J Hematol. 2015 Dec;90 Suppl 2:S3-10. doi: 10.1002/ajh.24220. PMID 26619194
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com